CLINICAL TRIAL: NCT01604811
Title: Exploratory Study of L.S.E.S.r. (PERMIXON® 160 mg Hard Capsule) Versus Tamsulosine LP Activity on Inflammation Biomarkers in the Treatment of Urinary Symptoms Related to BPH; a Multinational, Multicentric, Randomised, Double Blind Parallel-group Prospective Study
Brief Title: Exploratory Study of L.S.E.S.r. (LipidoSterolic Extract of Serenoa Repens)(PERMIXON® 160 mg Hard Capsule) Versus Tamsulosine LP Activity on Inflammation Biomarkers in Urinary Symptoms Related to BPH (Benign Prostatic Hyperplasia)
Acronym: PERMIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: P00048 GP 4 03; 2011-005307-33 (EudraCT Number)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-07

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — saw palmetto extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tested product (Experimental)
  Interventions: Drug: Permixon® 160 mg; Drug: Placebo matching Tamsulosine Arrow LP
- Comparator (Active Comparator)
  Interventions: Drug: Tamsulosine Arrow LP; Drug: Placebo matching Permixon® 160 mg

INTERVENTIONS:
Drug: Permixon® 160 mg — Oral administration - 160 mg twice daily.
  Arms: Tested product
Drug: Tamsulosine Arrow LP — Oral administration - 0.4 mg daily.
  Arms: Comparator
Drug: Placebo matching Permixon® 160 mg — Oral administration - twice daily.
  Arms: Comparator
Drug: Placebo matching Tamsulosine Arrow LP — Oral administration - daily.
  Arms: Tested product

SUMMARY:
Inflammation is reported as one of the most recent hypotheses to explain BPH. Recent published works pointed out that urine and serum markers could be used for detection of prostatic inflammation.

The aim of the study is to assess the activity on inflammation biomarkers (serum and urine inflammation markers) of Permixon® 160 mg hard capsule and Tamsulosine Arrow LP in the treatment of urinary symptoms related to BPH.

The potential links between serum and urinary markers of inflammation and BPH clinical symptoms at baseline and on treatment will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Between 45 and 85 years old.
* Patient with bothersome lower urinary tract symptoms such as pollakiuria (daytime or night time), urgency, sensation of incomplete voiding, delayed urination or weak stream, existing for over 12 months
* I-PSS ≥ 10 at selection visit and ≥ 12 at randomisation visit (visit 2)
* Stable patient's disease at randomisation defined as an absolute difference of 2 or less on I-PSS between selection and randomisation visits (visit 1 and visit 2)
* I-PSS QoL score ≥ 3 evaluated at selection and randomisation visits,
* 5 mL/s ≤ maximum urinary flow rate < 15 mL/s for a voided volume ≥ 150 mL and ≤ 500 mL evaluated at randomisation visit (2 measurements if necessary)
* Prostatic volume ≥30 cm³ determined by transrectal ultrasound at randomisation visit (visit 2)
* Serum total PSA at randomisation visit (visit 2) :

  * 4 ng/mL
  * 10 ng/mL and Prostate Specific Antigen (free) / Prostate Specific Antigen (total) ≥ 25% or negative prostate biopsy within the past 6 months prior to selection visit.
* Patient able to understand and sign the informed consent and understand and fill in self-questionnaires

Exclusion Criteria:

* Post-void residual urine volume > 200 mL (by suprapubic ultrasound) at randomisation visit (visit 2).
* Urological history :

  * Urethral stricture disease and/or bladder neck disease
  * Active (at selection and randomisation visits) or recent (< 3 months) or recurrent urinary tract infection
  * Indication of BPH surgery
  * Stone in bladder or urethra
  * Acute or chronic (documented) prostatitis
  * Prostate and cancer cancer treated or untreated
  * Interstitial cystitis (documented by symptoms and/or biopsy)
  * Active upper tract stone disease causing symptoms
* Patient with history of surgery of the prostate, bladder neck or pelvic region
* Any local and/or systemic inflammation disorders at selection and randomisation visit

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Inflammation Biomarkers | Day 1 (baseline), Day 30, Day 90
  "Inflammation biomarkers assay in patients suffering from Benign Prostatic Hyperplasia at Day 1, Day 30 and Day 90 :
  * Urine inflammation markers [mRNA (messenger RiboNucleic Acid) and proteins] on the first urine flow after digital rectal examination
  * Serum inflammation markers (C-Reactive Protein and Sedimentation Rate) "

SECONDARY OUTCOMES:
Change from baseline of urinary symptoms | Day 1 (baseline), Day 30, Day 90
  Urinary symptoms assessed by International Prostate Symptom Score (I-PSS) (self-administered questionnaire)
Change from baseline of quality of life | Day 1 (baseline), Day 30, Day 90
  Impact of symptoms on quality of life on the basis of the I-PSS quality of life question scored by the patient
Change from baseline of sexual activity | Day 1 (baseline), Day 30, Day 90
  Sexual activity assessed by the Male Sexual Function questionnaire (MSF-4) (self-administered questionnaire)
Change from baseline of maximum urinary flow rate | Day 1 (baseline), Day 30, Day 90
  Uroflowmetry performed using an electronic flow meter.
Change from baseline of prostate volume | Day 1 (baseline), Day 30, Day 90
  Prostate volume determined by transrectal ultrasound
Change from baseline of post-void residual urine volume (PVR) | Day 1 (baseline), Day 30, Day 90
  Post-void residual urine volume determined by suprapubic ultrasound.
Number of adverse events | up to 90 days
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (32):
- France (16):
  - Angers
  - Bordeaux
  - Cornebarrieu
  - Créteil
  - La Tronche
  - Le Fousseret
  - Limoges
  - Lyon
  - Marseille
  - Nice
  - Paris
  - Saint-Orens-de-Gameville
  - Segré
  - Seysses
  - Tiercé
  - Toulouse
- Italy (8):
  - Bari
  - Catanzaro
  - Florence
  - Genova
  - Milan
  - Perugia
  - Pisa
  - Trieste
- Portugal (2):
  - Lisbon
  - Porto
- Spain (6):
  - A.Coruna
  - Barcelona
  - Bilbao
  - Madrid
  - Sabadell
  - Seville